CLINICAL TRIAL: NCT07099157
Title: Efficacy and Safety of Brivudine in the Treatment of Herpes Zoster: A Multicenter, Randomized, Prospective Clinical Trial
Brief Title: Efficacy and Safety of Brivudine in the Treatment of Herpes Zoster
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Peking University Third Hospital (Other)
Collaborators: Peking University First Hospital (Other); Air Force Military Medical University, China (Other); Beijing Hospital of Traditional Chinese Medicine (Other); Xuanwu Hospital, Beijing (Other)
Responsible Party: Principal Investigator, Guo Jin-Zhu, Deputy Director of Dermatology, Peking University Third Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: M20250600
Record Dates: First submitted 2025-07-18; First posted 2025-08-01 (Actual); Last update posted 2026-01-02 (Actual); Status verified 2025-12

CONDITIONS: Herpes Zoster
Keywords: Herpes Zoster; Brivudine; pain; treatment
MeSH Terms: conditions — Herpes Zoster; Pain | interventions — brivudine; Famciclovir

STUDY DESIGN:
Intervention Model Description: Participants receive either Brivudine (125mg/day) or Famciclovir (dose-adjusted by creatinine clearance) for 7 days.
Who Masked: Investigator
Masking Description: Blinded Investigator conduct the follow-ups.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Brivudine Group (Experimental)
  Interventions: Drug: Brivudine
- Famciclovir Group (Active Comparator)
  Interventions: Drug: Famciclovir

INTERVENTIONS:
Drug: Brivudine — brivudine 125 mg per dose, once daily, 7 days
  Arms: Brivudine Group
Drug: Famciclovir — orally receive famciclovir at doses adjusted based on creatinine clearance (CrCl), 7 days
  Arms: Famciclovir Group

SUMMARY:
This multicenter RCT aims to compare the efficacy and safety of Brivudine versus Famciclovir in treating acute herpes zoster. Primary objective: Evaluate pain reduction via Numeric Pain Rating Scale (NPRS) at Day 30. Secondary objectives: Compare NPRS at Day 3/Day 7/Day 14/Day 90, time to lesion resolution, Postherpetic Neuralgia (PHN) incidence, and safety.

DETAILED DESCRIPTION:
A randomized controlled trial enrolling 140 participants from 5 centers in China. Patients receive either Brivudine (125mg/day) or Famciclovir (dose-adjusted by creatinine clearance) for 7 days. Follow-ups occur at Day 3, Day 7, Day 14, Day 30, Day 90. Primary endpoint: Numeric Pain Rating Scale (NPRS) at Day 30; secondary endpoints: NPRS at other timepoints, lesion healing time, Postherpetic Neuralgia (PHN) rate, and adverse events.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years, regardless of gender;
2. Signed Informed Consent Form;
3. Female subjects must not plan for pregnancy or oocyte donation from screening until 1 week after the last dose and must voluntarily adopt highly effective physical contraception; male subjects must not plan for fertility or sperm donation during the same period and must voluntarily adopt highly effective physical contraception. Methods include:

   * Barrier methods: Condom or barrier cap (diaphragm or cervical cap);
   * Intrauterine device (IUD) or intrauterine system (IUS);
   * Surgical sterilization (bilateral oophorectomy with/without hysterectomy, total hysterectomy, bilateral tubal ligation, or vasectomy) performed ≥6 months prior to the first dose in the subject or their partner;
   * Other investigator-confirmed highly effective physical contraception.

Exclusion Criteria:

1. Allergy to brivudine, famciclovir, or penciclovir;
2. Current use of fluorouracil agents (e.g., 5-fluorouracil, capecitabine, tegafur, flucytosine);
3. Cancer patients currently undergoing chemotherapy;
4. Pregnant or lactating women;
5. Parkinson's disease;
6. Any condition deemed inappropriate for study participation by the investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2025-08-25 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Day 30 numeric pain rating scale (NPRS) | Day 30
  Scores range from 0 to 10, where 0 represents no pain and 10 represents the worst pain imaginable. Higher scores indicate greater pain intensity.

SECONDARY OUTCOMES:
numeric pain rating scale (NPRS) on Day 3, Day 7, Day 14, Day 90 | Day 3, Day 7, Day 14, Day 90
  Scores range from 0 to 10, where 0 represents no pain and 10 represents the worst pain imaginable. Higher scores indicate greater pain intensity.
Incidence of PHN | Day 90
  Incidence of Postherpetic Neuralgia
skin lesion on Day 3, Day 7, Day 14, Day 30, Day 90 | Day 3, Day 7, Day 14, Day 30, Day 90
  whether the presence of hemorrhagic bullae, bullae, erosions, or ulcers
Lesion area on Day 3, Day 7, Day 14, Day 30 and Day 90 | Day 3, Day 7, Day 14, Day 30 and Day 90
  Percentage of body surface area (BSA%) affected by lesions on Day 3, Day 7, Day 14, Day 30 and Day 90
cessation of new lesion formation | Day 3, Day 7, Day 14, Day 30 and Day 90
  whether cessation of new papule/vesicle formation on Day 3, Day 7, Day 14, Day 30 and Day 90
complete crusting of all lesions | Day 3, Day 7, Day 14, Day 30 and Day 90
  whether complete crusting of all lesions Day 3, Day 7, Day 14, Day 30 and Day 90
Adverse Events (AEs) and Serious Adverse Events (SAEs) | From baseline to Day 30
  Adverse Events (AEs) and Serious Adverse Events (SAEs) in 30 days

CONTACTS AND LOCATIONS:
Locations (4):
- China (4):
  - Peking University Third Hospital, Beijing
  - Beijing Hospital of Traditional Chinese Medicine, Capital Medical University, Beijing
  - Peking University First Hospital, Beijing
  - Xuanwu Hospital, Capital Medical University, Beijing

IPD SHARING:
Plan to Share IPD: No